CLINICAL TRIAL: NCT07046728
Title: Observationnal Multicentric Study to Evaluate the Safety and the Efficacy of DAROMUN of Melanoma Patient (Resectable Stage IIIB to IIID) Treated by Intralesionnal Injection
Brief Title: Efficay and Safety of DAROMUN on Patient Treated by Intralesionnal Injection: DAROMEL
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Dermato01
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Injections Intralesional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Efficay and Safety of DAROMUN on patient treated by intralesionnal injection: DAROMEL — Observationnal study with clincal data collection to evaluate the efficiency and the tolerability of DAROMUN

SUMMARY:
Melanoma is a malignant tumor originating from melanocytes, with a high metastatic potential, particularly in advanced stages. The standard treatment for resectable melanomas has traditionally been surgery, often followed by adjuvant therapy to reduce the risk of recurrence. However, the emergence of neoadjuvant/perioperative therapies, administered prior to surgery, has revolutionized the management of patients with stage IIIB-C-D melanoma presenting with locoregional macroscopic metastases. Another therapeutic approach involving an intratumoral immunocytokine called DAROMUN (a fusion protein combining an antibody and a cytokine), designed to stimulate antitumor immunity within the melanoma cell microenvironment, was presented at the global oncology congress (ASCO) in June 2024. Preliminary biomarker analyses indicated that treatment with DAROMUN leads to an increase in tumor-infiltrating lymphocytes, particularly CD4+ and CD8+ cells, suggesting immune activation within the tumor microenvironment. This molecule, recently made available through a compassionate use program on the website of the French National Agency for the Safety of Medicines and Health Products (ANSM), may be particularly beneficial for patients who experience recurrence despite prior adjuvant therapy and who have locally advanced, resectable melanoma.The team therefore aim to conduct a real-world, ambispective, multicenter study under the auspices of the Cutaneous Oncology Group (GCC) of the French Society of Dermatology (SFD), focusing on the use of DAROMUN in patients with stage IIIB-IIID locally advanced melanoma.The primary endpoint will be to assess the response rate to treatment according to RECIST 1.1 criteria.Secondary endpoints will include: distant metastasis-free survival, pathological complete response rate, treatment safety profile, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old with locally advanced melanoma stage IIIB, IIIC, or IIID.
* Patient diagnosed with cutaneous melanoma or melanoma of unknown primary origin.
* Disease progression after treatment with immunotherapy in the adjuvant or metastatic setting.
* Patient having a contraindication to immunotherapy.
* Patient having received at least one intralesional infusion of Daromun.

Exclusion Criteria:

* Patient with uveal or mucosal melanoma.
* Opposition to data use (withdrawal of non-opposition).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate according to RECIST 1 ( Evaluation Criteria In Solid Tumors ) | From baseline to 13 months ( september 1, 2024 to october 31, 2025)
  Objective response rate according to RECIST 1 ( Evaluation Criteria In Solid Tumors )

SECONDARY OUTCOMES:
Pathological complete response rate (macroscopic) | From baseline to 13 months ( september 1, 2024 to october 31, 2025)
  Disappearance of the disease at the macroscopic levels
Pathological complete response rate (microscopic) | From baseline to 13 months ( september 1, 2024 to october 31, 2025)
  Disappearance of the disease at the microscopic levels

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nice, Nice, Alpes Maritimes, France